CLINICAL TRIAL: NCT01717690
Title: Randomized Controlled Clinical Trial of 2% Chlorhexidine Gluconate-Impregnated Bath Cloths to Prevent MRSA Colonization on Complex Continuing Care Units of Baycrest Hospital
Brief Title: Study of 2% Chlorhexidine Gluconate-Impregnated Bath Cloths to Prevent MRSA Colonization in Complex Continuing Care
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baycrest (Other)
Responsible Party: Principal Investigator, Chingiz Amirov, Director, Infection Prevention and Control, Baycrest
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BCGC-CHG-2012
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Staph Aureus Methicillin Resistant Colonization
Keywords: MRSA; chlorhexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHG antiseptic body cleanser (Active Comparator): One randomly selected intervention unit in Complex Continuing Care program where all patients (MRSA-positive and MRSA-negative) will be bathed daily with an antiseptic body cleanser (CHG).
  Only MRSA-negative patients at enrollment will be included in the study analysis, and only their outcomes (MRSA status and time to conversion) will be analyzed.
  Antiseptic body cleanser - 2% Chlorhexidine Gluconate in a non-alcohol and non-alkaline base, delivered to skin surface through the bath cloths impregnated with this antiseptic solution.
  Interventions: Drug: CHG antiseptic body cleanser
- Non-antiseptic body cleanser (No Intervention): Two control units in Complex Continuing Care program where all patients (MRSA-positive and MRSA-negative) will be bathed daily with a non-antiseptic body cleanser (Comfort Bath ®).
  Only MRSA-negative patients at enrollment will be included in the study analysis, and only their outcomes (MRSA status and time to conversion) will be analyzed.

INTERVENTIONS:
Drug: CHG antiseptic body cleanser — The intervention consists of daily bathing of all patients (MRSA-positive and MRSA-negative) on the intervention unit with CHG.
  Other Names: Chlorhexidine gluconate cloths; Drug Identification Number (Health Canada): 02245741
  Arms: CHG antiseptic body cleanser

SUMMARY:
The purpose of this study is to determine whether daily bathing with 2% chlorhexidine gluconate-impregnated antiseptic cleanser (CHG) significantly reduces incidence of colonization of hospitalized patients with methicillin-resistant Staphylococcus aureus (MRSA).

Investigators postulate that daily bathing with CHG significantly reduces incidence of colonization of hospitalized patients with MRSA.

DETAILED DESCRIPTION:
Bathing patients with 2% chlorhexidine gluconate-impregnated cloths (CHG) is an established practice at Baycrest. Our previous studies have demonstrated strong MRSA-preventive properties of CHG bathing practice - the rate of MRSA transmission on intervention units dropped from 4.99 to 0.88 cases per 1,000 patient days - an overall rate reduction of 82%.

Although CHG will continue to be used as part of an established clinical practice in our hospital, its impact on MRSA prevention merits further evaluation in complex continuing care (CCC) settings endemic for MRSA. Investigators propose a cluster-randomized, prospective, open-label, two-arm clinical trial (RCT) on three geographically separate, but otherwise comparable, CCC units - one intervention unit using CHG, and two control units using non-antiseptic cleanser. The RCT is expected to conclusively answer whether daily bathing with CHG significantly reduces incidence of MRSA colonization.

By cluster randomization investigators imply randomly assigning interventions to the three patient care units. Investigators propose randomization of the units as it is not feasible to randomly assign the individual participants to intervention vs control arms.

For a meaningful interpretation of the RCT findings, patient populations on the three floors will be compared at the beginning, during, and at the end of the study. The following variables will be used to compare patient populations:

* Colonization pressure (CP) is a measure of the MRSA reservoir on the unit. CP will be calculated at the onset of the RCT and then bi-weekly (Number of MRSA patient-days × 100 ÷ Total Number of Patient Days).
* Average Braden scale score (BSS) for patients on each unit is measured to predict a pressure ulcer risk. It is one of the measures of patient's clinical complexity. It is calculated by examining six patient criteria (sensory perception, skin moisture, physical activity, mobility, nutrition, friction and shear). BSS will be calculated at the onset of the RCT and then monthly.
* Average Case Mix Index (CMI) is a value reflecting the daily relative weight of resources used by an individual patient compared to a base resource level (the average resource use of the patient population). The CMI value is not a dollar amount; rather it is a relative value and an indirect marker of patient's clinical complexity. CMI will be calculated at the onset of the RCT and then quarterly.

Patient information will be de-identified for privacy reasons, before analysis of the study data - logistic regression, to compare the rates of MRSA incidence and time to MRSA conversion on intervention and control units.

ELIGIBILITY:
Inclusion Criteria:

* MRSA-negative (at enrollment) inpatient of Complex Continuing Care program

Exclusion Criteria:

* MRSA-positive (at enrollment) inpatient of Complex Continuing Care program

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2013-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Incidence of MRSA colonization | 12 months
  Primary outcome measure will be incidence of MRSA colonization measured through bi-weekly point-prevalence surveys on each of the three units. All new admissions and re-admissions to the units will also be screened. Protective properties of CHG bathing are expected to significantly reduce the incidence of MRSA transmission in the intervention arm, compared to control arms.

SECONDARY OUTCOMES:
Time to MRSA conversion | 12 months
  Secondary outcome measure will be time to MRSA conversion measured as the length of time it takes patients to convert from being MRSA-negative at enrollment to MRSA-positive at discharge or end of the study. Protective properties of CHG bathing are expected to significantly prolong conversion time.

CONTACTS AND LOCATIONS:
Overall Officials: Chingiz Amirov, MPH, CIC, Principal Investigator — Baycrest
Locations (1):
- Baycrest Hospital, Complex Continuing Care program, Toronto, Ontario, Canada